CLINICAL TRIAL: NCT00173095
Title: The Bilirubin Levels in Cerebrospinal Fluid of Spontaneous Subarachnoid Hemorrhage Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700413
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-01

CONDITIONS: Spontaneous Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
According to Morgan et. al. (J Neurosurg 101:1026-1029, 2004): bilirubin as a cerebrospinal fluid marker of sentinel subarachnoid hemorrhage: a preliminary report in pigs, we're going to test the hypothesis in the cerebrospinal fluid of spontaneous subarachnoid hemorrhage patients.

DETAILED DESCRIPTION:
According to Morgan et. al. (J Neurosurg 101:1026-1029, 2004): bilirubin as a cerebrospinal fluid marker of sentinel subarachnoid hemorrhage: a preliminary report in pigs, we're going to test the hypothesis in the cerebrospinal fluid of spontaneous subarachnoid hemorrhage patients. We'll collect the serial cerebrospinal fluid in 15-20 spontaneous subarachnoid hemorrhage patients to see the time sequence of changes in bilirubin levels.

ELIGIBILITY:
Inclusion Criteria:

* spontaneous subarachnoid hemorrhage in less than three days

Exclusion Criteria:

* spontaneous subarachnoid hemorrhage more than three days

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-01; Study Completion 2008-01

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Mu Chen, M.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taipei, Taiwan